CLINICAL TRIAL: NCT03773718
Title: Study of the Pathogenic Mechanisms of Metabolic Syndrome at the Background of Genetically Determined Insulin Resistance in Childhood Cancer Survivors
Brief Title: Metabolic Syndrome in Childhood Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: 0925-0586
Record Dates: First submitted 2018-12-07; First posted 2018-12-12 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; children; cancer; survivors; genetic
MeSH Terms: conditions — Metabolic Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Russkoe pole: 400 patients

SUMMARY:
The research is devoted to studying the features of the metabolic syndrome in cancer survivors in childhood is supposed to answer the following questions:

* How can metabolic syndrome be diagnosed in the Russian population of survivors of acute lymphoblastic leukemia and non-Hodgkin's lymphomas?
* What are the features of the clinical symptoms of metabolic syndrome in this category of patients?
* Which genetic mutations are found in cancer survivors of patients with metabolic syndrome; Which of these mutations can be considered as protective or vice versa predisposing to the development of metabolic syndromes? Is the metabolic syndrome associated with an increased frequency of toxic complications of therapy during the intensive stages?

DETAILED DESCRIPTION:
Brief Overview:

The remarkable progress in developing curative therapy for childhood cancer over the last 4 to 5 decades has increased awareness of the serious cancer treatment-related late effects experienced by long-term survivors such as premature mortality early deaths, second primary cancers, organ dysfunction (heart, lung, endocrine system), fertility impairment, cognitive deficits, and reduced quality of life. Endocrine disorders, which occur in 30% to 70% of childhood cancer survivors, are among the most frequent late effects of anticancer therapy. Survivors treated with radiation and alkylating agent chemotherapy for hematological malignancies and CNS tumors are at a particularly high risk for endocrine dysfunction.

Most anticancer drugs act directly or indirectly by modifying intracellular metabolism. Therefore, high frequency of acute and late cancer treatment-related organ toxicity can result in metabolic disorders. For example, steroid-induced hypercortism blocks glycolysis and results in insulin resistance of tissues. Insulin resistance is associated with earlier manifestation of diabetes mellitus, obesity etc. The clinical sequelae of metabolic syndrome developing in childhood cancer survivors may include insulin resistance, fasting hyperglycemia, endothelial failure, obesity, dyslipidemia, hypertension, chronic fatigue syndrome, motor and behavioral disorders.

Modern genetics make it possible to create a basis for a personalized approach to the prevention of early and late toxic effects caused by anticancer therapy and the rehabilitation of the childhood cancer survivors.

Objectives:

Specific Aim 1. Evaluate the frequency and clinical features of the metabolic syndrome in childhood cancer survivors.

Hypothesis 1A: Components of the metabolic syndrome are realizing in children and adolescents at all stages of therapy of leukemia and lymphomas, can influence the development of complications and late toxic effects.

Hypothesis 1B: Initial health conditions (abnormal IBM, family history, comorbid diseases); drug's toxicity could influence to the appearance of early manifestation of metabolic syndrome.

Specific Aim 2: Evaluate the contribution of functional polymorphisms in candidate genes to metabolic syndrome outcomes among childhood cancer patients.

Hypothesis 2A: Genetic polymorphisms involved in the regulation of the insulin resistance and cancer medications during treatment contribute to the development of metabolic syndrome in childhood cancer survivors.

Specific Aim 3: Assess the extent to which genetic predictors, doses of drugs, risk factors improve the discriminatory performance of standard clinical prediction models for metabolic syndrome outcomes among childhood cancer survivors.

Hypothesis 3 A: Development of metabolic syndrome in cancer patients depends of genetic determinants and toxic effects of antitumor therapy.

Secondary Aim 1: Assess the definition of metabolic syndrome in cohort of patients of leukemia and lymphoma and survivors.

Hypothesis 1A: Episodes of triglyceridemic, insulin resistance (Hyperglycemia, HOMA>2,7, Steroid Diabetes) during the treatment could be the base evidence marker of Metabolic Syndrome in patients treated by antitumor therapy.

Hypothesis 1 B: Endothelial dysfunction as a clinical component of metabolic syndrome is responsible for cardiovascular abnormalities in cancer survivors.

Exploratory Aim 1: Assess the association of biomarkers and genetic predictors among childhood cancer survivors with therapeutic exposures (chemotherapy and/or radiation therapy) and metabolic syndrome.

Evaluation:

Eligible persons who consent to participate in this trial will be asked to do the following:

* Vital sign measurement including resting heart rate, blood pressure, height, and weight.
* A total of 12 mL of blood will be collected in 3 test tubes. Biomarker analysis will be completed by Laboratory of Dmitry Rogachev National Medical Research Center.
* A Total of 4 mL of blood in 1 test tube will be used for genotyping for the presence of polymorphic variants in genes involved in the biotransformation of xenobiotics, insulin resistance and carbohydrate metabolism in the biomolecular laboratory of Dmitry Rogachev National Medical Research Center.
* An echocardiogram and ultrasound will be performed to assess cardiac function.
* CAVI and ABI pulse wave velocity will be non-invasively measured by using the SphygmoCor VaSera VS-1500N. Arterial pressure waveforms will be recorded with a strain gauge pressure sensor placed lightly over the radial artery before and after "6-minutes physical activity".

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors:
* Treatment with chemotherapy and/or radiation therapy for a primary ALL/NHL diagnosed prior to age 17 years.
* ≤ 15 years of age at the time of enrollment.
* No cytostatic drugs uptake during the study.

Exclusion Criteria:

* Diagnosis of diabetes mellitus types 1 or 2 types before antitumor therapy
* Active oncological disease
* History of allogeneic hematopoietic cell transplant
* The renouncement of participation from the patient or legally authorized representative

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants for this study will be patients of "Russkoe Pole" cohort, the study designed to evaluate health among children and adolescents survivors of childhood leukemia and lymphoma as they age. Participants in RPC undergo risk-based medical screening according to the Standards of Medical Insurance for rehabilitation of Cancer treated patients.
  To be eligible for RPC, cancer survivors must has been treated at Russian children oncology clinics by MB-ALL/ BFM-NHL and be 17 years of age or younger, and at least 6 months from the completion of the therapy. All the patients will has exhaustively full epicrisis of medical history with cumulative doses of medications. coz RPC is a retrospective cohort study with ongoing recruitment (additional survivors become eligible over time).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
The frequency of metabolic syndrome | 12 months
  The frequency of diagnosed metabolic syndrome in the cohort of children and adolescents with leukemia and lymphomas

SECONDARY OUTCOMES:
Genetic risk | 12 months
  The detection of NSP associated with metabolic syndrome in children and adolescents after childhood cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M. Hudson, MD, Study Chair — St. Jude Children's Research Hospital Memphis, TN 38105
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03773718/Prot_001.pdf